CLINICAL TRIAL: NCT05524272
Title: Stress-Relieving Effects of Colour-By-Number Mandalas ın Children Hospitalised Due to A Chronic Disease
Brief Title: Effects of Colour-By-Number Mandalas ın Children Hospitalised Due to A Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, DİDEM COŞKUN ŞİMŞEK, Principal Investigator, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Colour-By-Number Mandalas
Record Dates: First submitted 2022-02-14; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Child, Only; Chronic Diseases in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THE EFFECTS OF COLOUR BY NUMBER MANDALA (Experimental): This study was conducted to find out the effects of colour by number mandala in decreasing the stress of hospitalized children with chronic disease. A randomized controlled study.This study was conducted with 120 children between the ages of 8 and 11. 60 children formed the experimental group, while 60 children formed the control group. Descriptive Information Form and Perceived Stress Scale were used in data collection.
  Interventions: Other: This study aims to evaluate the effects of colour by number mandala in decreasing the stress of children hospitalized due to their chronic disease.

INTERVENTIONS:
Other: This study aims to evaluate the effects of colour by number mandala in decreasing the stress of children hospitalized due to their chronic disease. — Colour by number Mandala in different sizes includes pictures and numbers. The child has to find the colour specified in the number and colour it with the specified colour. Colourful pictures emerge as a result of colouring

SUMMARY:
Purpose: This study was conducted to find out the effects of colour by number mandala in decreasing the stress of hospitalized children with chronic disease.

Design: A randomized controlled study. Methods: This study was conducted with 120 children between the ages of 8 and 11. 60 children formed the experimental group, while 60 children formed the control group. Descriptive Information Form and Perceived Stress Scale were used in data collection.

DETAILED DESCRIPTION:
Experimental group: The children, along with their parents, were interviewed by one of the researchers on their first day of hospitalisation. The parents were informed about the Descriptive Information Form and the Perceived Stress Scale for Children, which the researcher filled out in the presence of the children and their parents. The children were then given a colour-by-number mandala and colouring pencils. A different colour-by-number mandala was given to each participant every day; the mean length of hospital stay was 3 days. At the end of the third day, the same researcher interviewed the children and filled out again the Perceived Stress Scale for Children.

ELIGIBILITY:
Inclusion Criteria:

* parents who agreed to participate in the study

Exclusion Criteria:

* visually impaired child
* mentally retarded child
* speech impaired children

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
this study was measured colour-by-number mandalas do reduce the perceived stress levels in children hospitalised due to a chronic disease. | 3 days
  A different colour-by-number mandala was given to each participant every day; the mean length of hospital stay was 3 days. At the end of the third day, the same researcher interviewed the children and filled out again the Perceived Stress Scale for Children.
  The Perceived Stress Scale for Children: A minimum of 0 and a maximum of 27 points are obtained from the scale. A high score from the scale indicates a high level of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat University, Elâzığ, Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No